CLINICAL TRIAL: NCT03975933
Title: Pregnancy Testing in Northern Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Ichuli Consulting Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UIUC_PT
Record Dates: First submitted 2018-07-30; First posted 2019-06-05 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-01

CONDITIONS: Pregnancy Tests
Keywords: Reproductive Health; Family Planning; Randomization Trial; Uganda
MeSH Terms: interventions — Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Free pregnancy tests at baseline but not for the future (Experimental): We offer free pregnancy test service at baseline but the respondents do not have an opportunity to receive or buy a pregnancy test.
  Interventions: Diagnostic Test: Pregnancy test at Baseline
- Free pregnancy tests at baseline and for the future (Experimental): We offer free pregnancy test service at baseline and a free pregnancy test for future use.
  Interventions: Diagnostic Test: Pregnancy test at Baseline; Diagnostic Test: Free pregnancy test for the future use
- Free pregnancy tests at baseline and future use (random price) (Experimental): We offer free pregnancy test service at baseline and the respondents have an opportunity to buy a pregnancy test.
  Interventions: Diagnostic Test: Pregnancy test at Baseline; Diagnostic Test: Pregnancy test for the future use with randomzied price
- Control Group (No Intervention): Control group. No intervention is implemented.
- Pregnancy test for the future use (Experimental): No free pregnancy tests at baseline, but receive a free pregnancy test for the future.
  Interventions: Diagnostic Test: Free pregnancy test for the future use
- Pregnancy test for the future with random price (Experimental): No free pregnancy tests at baseline, but receive an opportunity to buy a pregnancy test for the future (ranodmized price).
  Interventions: Diagnostic Test: Pregnancy test for the future use with randomzied price

INTERVENTIONS:
Diagnostic Test: Pregnancy test at Baseline — Among respondents who are randomly selected to receive a free home pregnancy test service, they will be offered the chance to take the test in the presence of the enumerator. Specifically, this would mean they would be given a cup to collect a sample of urine. The respondent would do so privately, then bring the cup back to the enumerator who would dip the home pregnancy tests and assist with interpreting the result. However, respondents can decline to take the test with the enumerator. Treatment assignment will be stratified by whether respondent use modern family planning at baseline.
  Arms: Free pregnancy tests at baseline and for the future; Free pregnancy tests at baseline and future use (random price); Free pregnancy tests at baseline but not for the future
Diagnostic Test: Free pregnancy test for the future use — We will provide a free pregnancy test in for the future use.
  Arms: Free pregnancy tests at baseline and for the future; Pregnancy test for the future use
Diagnostic Test: Pregnancy test for the future use with randomzied price — We will provide an opportunity to buy a pregnancy test for the future use with randomized price.
  Arms: Free pregnancy tests at baseline and future use (random price); Pregnancy test for the future with random price

SUMMARY:
Given the high rate of delayed adoption of antenatal care (ANC), and high rates of unintended pregnancy and unsafe abortion in Uganda, research on the period of time before confirmation of pregnancy is critical to understand underlying beliefs that guide behaviors ultimately important for maternal and neonatal health (UDHS, 2011; Hussain, 2013).

Home pregnancy tests - which now cost less than 10 cents each - have the potential to facilitate FP uptake and significantly improve reproductive, maternal and child health outcomes in sub-Saharan Africa, including Uganda. These tests are easy to administer, disposable, inexpensive, and have a low false positive rate. Yet, for women living in rural areas in sub-Saharan countries, these tests are typically unavailable outside of health centers or they are prohibitively expensive.

This study will investigate women's underlying beliefs about pregnancy status and examine how providing access to home-based pregnancy tests - thus facilitating earlier resolution of uncertainty of pregnancy status - influences such beliefs and decisions to take up family planning (FP).

The results will inform the design of a larger study in the future.

DETAILED DESCRIPTION:
Given the high rate of delayed adoption of antenatal care (ANC), and high rates of unintended pregnancy and unsafe abortion in Uganda, research on the period of time before confirmation of pregnancy is critical to understand underlying beliefs that guide behaviors ultimately important for maternal and neonatal health (UDHS, 2011; Hussain, 2013).

Unmet demand for contraceptives remains high in sub-Saharan Africa, with 25% of married women reporting wanting to avoid pregnancy but not currently using modern contraceptives (Clifton and Kaneda, 2013). One factor contributing to unmet demand is that women are refused access to hormonal contraceptives in some settings, because FP providers cannot rule out pregnancy if the woman is not menstruating at the time of her visit (Campbell et al., 2006; Shelton et al., 1992; Stanback et al., 1997). While the current standard is for health providers to use a simple six-question checklist to rule out pregnancy, the checklist has a false positive rate ranging from 11% to 64% (Tepper et al. 2013) and health workers often end up not trusting it (Comfort et al., 2016; Hoke et al., 2012). Pregnancy tests can give non-menstruating women the ability to confirm they are not pregnant and access hormonal contraceptive methods when they may otherwise be denied (Stanback et al., 2013). Greater access to pregnancy tests may also motivate women who are uncertain about their pregnancy status to adopt FP methods if they receive a negative test result and do not wish to have additional children. The administration of a home pregnancy test by a FP provider, including community health workers, can also serve as an opportunity for FP counseling which may further increase uptake.

Confirmation of negative pregnancy status can also reduce psychological anxiety, especially for women who may wish to delay or avoid becoming pregnant. Among women who may be using different forms of contraceptives, confirmation of negative pregnancy could provide proof of the methods' effectiveness thereby encouraging these women to continue use. Almost half of women in Uganda who adopt a contraceptive method discontinue use within 12 months and about 13% discontinue use of short-acting hormonal contraceptives because of method failure ((UBOS) and International 2012). Especially among women using these particular methods, confirming their negative pregnancy status could encourage them to continue use. For women with partners who want to delay or avoid pregnancy, confirming negative pregnancy status could reduce domestic violence and reduce marital distress. In Uganda, almost 60% of women have experienced physical violence in their lifetime, and 60% of these women report that perpetrator was their current spouse ((UBOS) and International 2012). In addition, among Ugandan women who have ever been pregnant, 16% report having experienced physical violence during pregnancy; the likelihood of violence during pregnancy is higher for women who have five or more children, lower education, or lower income ((UBOS) and International 2012). Confirmation of negative pregnancy could also aid with household decision-making and planning; for example, women who confirm they are not pregnant could make greater investment (financial, time, physical) in their children.

Although coverage for at least one ANC visit is high in most developing countries, this is not predictive of coverage for at least four visits - the previous number of recommended visit by the World Health Organization (AbouZahr and Wardlaw, 2001) and is far from reaching the most recent WHO recommendation of at least 8 visits during a pregnancy (WHO 2016). According to the 2011 Uganda Demographic and Health Survey, 95% of women receive ANC from a skilled provider. However, only 48% attend four or more visits, and the median gestational age at the first visit is 5.1 months - well into the second trimester - even though the WHO recommends initiating ANC as early as possible (UDHS, 2011). There is some existing evidence suggesting that women wait to seek ANC because of uncertainty about their pregnancy status (Myer and Harrison, 2003).

In addition, earlier recognition of a pregnancy could allow women to plan for unwanted pregnancies. For pregnancies that are carried to term, earlier recognition would allow women to adopt healthy prenatal behaviors earlier (such as avoiding alcohol consumption and smoking, taking prenatal vitamins, and using antimalarial bednets). Women would be better able to plan for the delivery, including saving for delivery-related costs, such as transportation, provider fees, and facility fees and planning for the location of the delivery and attendance at delivery. It would also allow women to adopt effective malaria prevention behaviors; while the WHO recommends that pregnant women receive intermittent preventive treatment for malaria as soon as possible in the 2nd trimester, pregnant women should be using anti-malarial bednets during the 1st trimester (when iPTP is contra-indicated) to protect against malaria infection, which can result in maternal and fetal anemia, placental parasitaemia, low birth weight, and neonatal mortality (WHO 2012).

Home pregnancy tests - which now cost less than 10 cents each - have the potential to facilitate FP uptake and significantly improve reproductive, maternal and child health outcomes in sub-Saharan Africa, including Uganda. These tests are easy to administer, disposable, inexpensive, and have a low false positive rate. Yet, for women living in rural areas in sub-Saharan countries, these tests are typically unavailable outside of health centers or they are prohibitively expensive. This study will investigate women's underlying beliefs about pregnancy status and examine how providing access to home-based pregnancy tests - thus facilitating earlier resolution of uncertainty of pregnancy status - influences such beliefs and decisions to take up family planning (FP) or seek appropriate pregnancy services.

This protocol outlines our proposed study. The results will inform the design of a larger study.

a. Objectives

The main objectives of this study are to understand the impact of increasing women's access to home pregnancy tests on reproductive health care seeking. In this study we focus on non-pregnant women and subsequent effects of access to pregnancy tests. Specifically, the main research questions of the proposed study are:

1. Beliefs: How do women form their beliefs about their pregnancy status, risk of pregnancy and how do these beliefs correlate with behaviors related to contraceptive adoption among non-pregnant women?
2. Effects of access to pregnancy tests: What are the effects of resolving uncertainty through home pregnancy tests on beliefs and reproductive behaviors including FP uptake, psychological well-being, and contraceptive continuation)?
3. Demand/Value of pregnancy tests: What is take-up of free pregnancy tests and if the test is distributed for free, at what point in time in the month (in relationship to their menstrual cycle or sexual behavior) do women most value using it if they are distributed for free? Does willingness to pay for these tests vary by prior experience with pregnancy tests and key characteristics such as age and number of previous pregnancies?

We hypothesize that providing access to pregnancy tests could influence reproductive behaviors in the following ways:

Hypothesis 1: For women who test negative, confirmation of negative pregnancy status using home pregnancy tests will facilitate adoption of modern contraceptives to prevent unintended pregnancies and reduce anxiety.

Hypothesis 2: Women who are most uncertain of their pregnancy status (correlated with beliefs and sexual behavior) will have a higher value of the pregnancy test (more willing to adopt or higher willingness to pay).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35
* Live in the catchment area
* Sexually Active

Exclusion Criteria:

* Currently, pregnant women or women who recently gave birth (within 6 weeks of interview)
* Already using long-term family planning methods (IUD, implant, sterilization)

End Survey if

* Women in menopause
* Women with sterilization
* Women with husband/partner with sterilization
* Women with long-term family planning methods (IUD and implant)
* Women who do not understand what menstrual period is
* Women who is currently pregnant or who recently gave a birth (within 6 weeks of interview)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1033 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Binary measures for the family planning take up | 1 month after baseline
  Use of short-term modern family planning short-acting reversible methods. We will measure take up as binary variables.
Binary measure of purchase of pregnancy test kit by price | 1 month after baseline
  Binary measures for the purchase of pregnancy test kit after baseline. Demand for pregnancy test kit is computed by Take it or leave it (TIOLI) method.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Thornton, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Ichuli Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamei A, Sato R, Thornton R. Factors associated with knowledge and use of home pregnancy test kits in Uganda. PLOS Glob Public Health. 2023 Jul 13;3(7):e0002165. doi: 10.1371/journal.pgph.0002165. eCollection 2023. PMID 37440465
- [Derived] Kamei A, Sato R, Thornton R. Effect of pregnancy tests on demand for family planning: evidence from a randomized controlled trial in Uganda. Reprod Health. 2021 Nov 15;18(1):231. doi: 10.1186/s12978-021-01279-5. PMID 34781969